CLINICAL TRIAL: NCT01154777
Title: COLLABORATIVE STUDY OF NEUROFEEDBACK TRAINING OF 6-18YEAR OLDS WITH AUTISM
Brief Title: Collaborative Study Of Neurofeedback Training Of 6-18 Year Olds With Autism
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute for Personal Excellence, P.A. (Other)
Collaborators: Life Quality Resources (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Magdalena M. Gebska-Wojdynska, M.D., Institute for Personal Excellence, P.A
Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NFB6-18Autism
Record Dates: First submitted 2010-06-29; First posted 2010-07-01 (Estimated); Last update posted 2010-10-05 (Estimated); Status verified 2010-10

CONDITIONS: Autism
Keywords: Neurofeedback; Braintraining; Autism; Mild; Moderate; Mild to Moderate Autism
MeSH Terms: conditions — Autistic Disorder; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Neurofeedback training — 60 sessions of Neurofeedback on 6-18 year olds with Autism

SUMMARY:
Neurofeedback, a neuro-cognitive training method based on operant conditioning, will be employed with 90 children with the Autistic Spectrum Disorders (ASD) over a 60 session training period to improve the limiting behavioral and sensory symptoms Autism presents (with each collaborative site working with 45 of the 90 participants). This study seeks to demonstrate that Neurofeedback training, a non-invasive approach based on Learning Theory, will mitigate presenting symptoms of Autism, and ultimately render the person with Autism significantly more able to interact with his/her environment successfully, independently function on a day-to-day basis, and improve overall mental health.

DETAILED DESCRIPTION:
The specific objective is to demonstrate quantitative and qualitative improvements in functional and behavioral parameters in individuals affected by Autism Spectrum Disorders when 60 Neurofeedback training sessions are applied. The long term objectives for these individuals include improvement of quality of daily functioning, better ability to integrate and navigate within society, and overall to decrease the limitations caused by the disability. Additionally, increasing awareness by the public, as well as healthcare providers and legislation, that Neurofeedback is a viable intervention which may contribute not only to a significant reduction of the level of disability for affected individuals, but also in reducing required lifetime costs of healthcare. Hopefully in the future Neurofeedback training would be incorporated as a standard of care for ASD. As of today, there are around 1000 trained Neurofeedback practitioners in the US who are offering this intervention to a very limited number of individuals due to lack of recognition of NFB benefits.

ELIGIBILITY:
Inclusion Criteria:

* 6 to 18 year olds who have been diagnosed by their physician with mild to moderate autism, in accordance with DSM-IV diagnostic criteria

Exclusion Criteria:

* Any child with a diagnosis of Bipolar Disorder, Tourette's Syndrome, an uncontrolled seizure disorder, or a history of any major psychiatric disorder will be excluded from eligibility for the study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-07; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Level of normalization of brainwaves based upon QEEG | Pre - training, 20 and 40 Session Interims, and post-training
  After completion of all neurofeedback sessions, post-training evaluation will include cognitive testing, completion of ASRS and ATEC forms and a post-QEEG. Interviews with parents will also be conducted to identify progress and changes in symptom presentation.

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena M Gebska-Wojdynska, M.D., Principal Investigator — Institute for Personal Excellence, P.A.; Lucy Chartier, Ph.D., NP, Principal Investigator — Life Quality Resources
Locations (2):
- United States (2):
  - Institute for Personal Excellence, P.A., Raleigh, North Carolina
  - Life Quality Resources, Raleigh, North Carolina

REFERENCES:
- See also: Life Quality Resources — http://www.lifequalityresources.org